CLINICAL TRIAL: NCT06726460
Title: Validation of the Accuracy of a Novel POCT Dry Electrolyte Analysis System in the Acute Care Setting: A Cross-Sectional Study
Brief Title: Validation of the Accuracy of a Novel POCT Dry Electrolyte Analysis System in the Acute Care Setting
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KY-405-01
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Electrolyte Disorder; Arrhythmia; Stroke
Keywords: Electrolyte Analyzer; Accuracy; P1; Eaglenos
MeSH Terms: conditions — Arrhythmias, Cardiac; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The biospecimens to be retained in this study will include serum and whole blood samples. The serum samples are residual specimens collected after electrolyte testing on an automated biochemical analyzer in the laboratory. These samples will be tested for electrolytes on both the Nova blood gas analyzer and the novel POCT dry electrolyte analysis system (P1) simultaneously. The whole blood samples are residual specimens collected after other blood tests are performed on the Nova system. These samples will also be tested for electrolytes on both the Nova system and P1 simultaneously.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Nova Group: This group involves the use of the Nova Stat Profile pHOx Ultra Analyzer System for measuring serum and whole blood samples. The results obtained from Nova will be compared with those obtained from P1.
  Interventions: Diagnostic Test: Nova Stat Profile pHOx Ultra Analyzer System(Nova)
- Group 1: P1 Group: This group involves the use of the novel POCT dry electrolyte analysis system P1 for measuring serum and whole blood samples. The results obtained from P1 will be compared with those obtained from Nova.
  Interventions: Diagnostic Test: Novel POCT dry electrolyte analysis system(P1)

INTERVENTIONS:
Diagnostic Test: Nova Stat Profile pHOx Ultra Analyzer System(Nova) — This group involves the use of Nova for measuring serum and whole blood samples. The results from Nova will be compared with those obtained from P1.
  Groups: Group 1: Nova Group
Diagnostic Test: Novel POCT dry electrolyte analysis system(P1) — This group involves the use of P1 for measuring serum and whole blood samples. The results from P1 will be compared with those obtained from Nova.
  Groups: Group 1: P1 Group

SUMMARY:
The goal of this study is to compare the performance of a novel Point-of-Care Testing (POCT) dry electrolyte analyzer (P1) with the Nova Stat Profile pHOx Ultra Analyzer System (Nova) in an acute care setting. The main questions it aims to answer are:

1. How consistent are the results between P1 and Nova in the emergency setting, including outliers, correlation, linearity, and bias?
2. Whether P1 can serve as a suitable alternative to Nova in the acute care setting for electrolyte measurement in the emergency environment.

Participants will be patients in the emergency department who will undergo simultaneous measurement with P1 and Nova during their emergency care to assess the performance of both devices.

Additionally, the study will investigate electrolyte levels in emergency patients, focusing on the prevalence of abnormal ionized magnesium (iMg2+) levels, the correlation between iMg2+ and total magnesium (tMg), and the clinical significance of iMg2+ measurement.

DETAILED DESCRIPTION:
This observational study aims to compare the performance of two electrolyte analysis systems, the electrolyte analyzer P1 and the Nova Stat Profile pHOx Ultra Analyzer System, in an emergency department (ED) or emergency intensive care unit (ICU) setting. The study will evaluate the consistency, correlation, and bias between the two electrolyte analysis systems. The study design is observational, with no intervention or treatment assigned to the participants. The comparison will be made using residual blood samples collected as part of routine care, following standard clinical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo electrolyte measuring in the emergency department (ED) or emergency intensive care unit (ICU).

Exclusion Criteria:

* Patients with a confirmed history of infectious diseases such as hepatitis B, syphilis, HIV/AIDS, etc.
* Missing residual sample types (serum or whole blood).
* Patients whose residual blood samples are not tested within the specified time frame after collection.
* Other patients deemed ineligible by the investigator.

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients presenting to the emergency department (ED) or admitted to the emergency intensive care unit (ICU) who are scheduled to undergo electrolyte measuring.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Consistency between P1 and Nova system for electrolyte parameters. | Within 30 minutes of serum sample collection and within 1 minute of whole blood sample collection
  This outcome measure is to evaluate the consistency between the novel POCT dry electrolyte analysis system (P1) and the Nova Stat Profile pHOx Ultra Analyzer System (Nova). Consistency will be assessed by comparing the results of electrolyte parameters (e.g., Sodium (Na+), Potassium (K+), Chloride (Cl-), Ionized calcium (iCa2+), Ionized magnesium (iMg2+)) and will be evaluated using Bland-Altman analysis.
Correlation between P1 and Nova for electrolyte parameters. | Within 30 minutes of serum sample collection and within 1 minute of whole blood sample collection
  This outcome measures the correlation between P1 and Nova for electrolyte parameters (e.g., Na+, K+, Cl-, iCa2+, iMg2+). The correlation will be quantified using Pearson's correlation coefficient
Bias at clinical decision levels between P1 and Nova. | Within 30 minutes of serum sample collection and within 1 minute of whole blood sample collection
  This outcome measure is to evaluate the bias at clinical decision levels between P1 and Nova. Bias will be assessed by calculating the difference in the results of key electrolyte parameters (e.g., Na+, K+, Cl-, iCa2+, iMg2+) between the two analysis system at clinically relevant thresholds. These thresholds will be based on established clinical decision points where treatment decisions are made.
Outlier Detection in electrolyte Parameters | Within 30 minutes of serum sample collection and within 1 minute of whole blood sample collection
  This outcome measure aims to identify and evaluate outliers in the electrolyte parameters measured by P1 and Nova. Outliers will be detected using statistical methods such as the Grubbs test or the Interquartile Range (IQR) method. The impact of these outliers on the consistency and accuracy of the measurements will also be assessed.

SECONDARY OUTCOMES:
Prevalence of abnormal iMg2+ (ionized magnesium) levels in emergency patients. | Within 30 minutes of serum sample collection and within 1 minute of whole blood sample collection
  This outcome will assess the prevalence of abnormal ionized magnesium (iMg2+) levels in patients admitted to the emergency department or emergency ICU.
Correlation between iMg2+ (ionized magnesium) and tMg (total magnesium) levels. | Within 30 minutes of serum sample collection
  This outcome will evaluate the correlation between ionized magnesium (iMg2+) levels and total magnesium (tMg) levels, with tMg levels obtained from central laboratory test results, in emergency patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Xie, Principal Investigator — Zhujiang Hospital, Southern Medical University Organization
Locations (1):
- Zhujiang Hospital, Southern Medical University Organization, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Data will be made available to qualified researchers upon submission of a research proposal and execution of a data use agreement. Data access will be granted after the final study results are published and after an ethical review by the institution's ethics board. Data sharing will be coordinated via email. Qualified researchers can contact zjyyllxs@126.com to request access to the data.

REFERENCES:
- [Background] Khan AI, Pratumvinit B, Jacobs E, Kost GJ, Kary H, Balla J, Shaw J, Milevoj Kopcinovic L, Vaubourdolle M, Oliver P, Jarvis PRE, Pamidi P, Erasmus RT, O'Kelly R, Musaad S, Sandberg S. Point-of-care testing performed by healthcare professionals outside the hospital setting: consensus based recommendations from the IFCC Committee on Point-of-Care Testing (IFCC C-POCT). Clin Chem Lab Med. 2023 Jun 2;61(9):1572-1579. doi: 10.1515/cclm-2023-0502. Print 2023 Aug 28. PMID 37267483
- [Background] Shi Q, Ba G, Li K, Mao Z. Is it practical to incorporate point-of-care testing into clinical prediction models for emergency? Intern Emerg Med. 2023 Oct;18(7):2155-2156. doi: 10.1007/s11739-023-03333-5. Epub 2023 Jun 6. No abstract available. PMID 37278909
- [Background] Johansson M, Whiss PA. Weak relationship between ionized and total magnesium in serum of patients requiring magnesium status. Biol Trace Elem Res. 2007 Jan;115(1):13-21. doi: 10.1385/BTER:115:1:13. PMID 17406070
- [Background] Escuela MP, Guerra M, Anon JM, Martinez-Vizcaino V, Zapatero MD, Garcia-Jalon A, Celaya S. Total and ionized serum magnesium in critically ill patients. Intensive Care Med. 2005 Jan;31(1):151-6. doi: 10.1007/s00134-004-2508-x. Epub 2004 Dec 17. PMID 15605229
- [Background] Oost LJ, van der Heijden AAWA, Vermeulen EA, Bos C, Elders PJM, Slieker RC, Kurstjens S, van Berkel M, Hoenderop JGJ, Tack CJ, Beulens JWJ, de Baaij JHF. Serum Magnesium Is Inversely Associated With Heart Failure, Atrial Fibrillation, and Microvascular Complications in Type 2 Diabetes. Diabetes Care. 2021 Aug;44(8):1757-1765. doi: 10.2337/dc21-0236. Epub 2021 Jun 18. PMID 34385344
- [Background] Rios FJ, Zou ZG, Harvey AP, Harvey KY, Nosalski R, Anyfanti P, Camargo LL, Lacchini S, Ryazanov AG, Ryazanova L, McGrath S, Guzik TJ, Goodyear CS, Montezano AC, Touyz RM. Chanzyme TRPM7 protects against cardiovascular inflammation and fibrosis. Cardiovasc Res. 2020 Mar 1;116(3):721-735. doi: 10.1093/cvr/cvz164. PMID 31250885
- [Background] Yogi A, Callera GE, Antunes TT, Tostes RC, Touyz RM. Transient receptor potential melastatin 7 (TRPM7) cation channels, magnesium and the vascular system in hypertension. Circ J. 2011;75(2):237-45. doi: 10.1253/circj.cj-10-1021. Epub 2010 Dec 7. PMID 21150127
- [Background] de Baaij JH, Hoenderop JG, Bindels RJ. Magnesium in man: implications for health and disease. Physiol Rev. 2015 Jan;95(1):1-46. doi: 10.1152/physrev.00012.2014. PMID 25540137
- [Background] Ye L, Zhang C, Duan Q, Shao Y, Zhou J. Association of Magnesium Depletion Score With Cardiovascular Disease and Its Association With Longitudinal Mortality in Patients With Cardiovascular Disease. J Am Heart Assoc. 2023 Sep 19;12(18):e030077. doi: 10.1161/JAHA.123.030077. Epub 2023 Sep 8. PMID 37681518
- [Background] Glasdam SM, Glasdam S, Peters GH. The Importance of Magnesium in the Human Body: A Systematic Literature Review. Adv Clin Chem. 2016;73:169-93. doi: 10.1016/bs.acc.2015.10.002. Epub 2016 Jan 13. PMID 26975973
- [Background] Olsson K, Ohlin B, Melander O. Epidemiology and characteristics of hyponatremia in the emergency department. Eur J Intern Med. 2013 Mar;24(2):110-6. doi: 10.1016/j.ejim.2012.10.014. Epub 2012 Nov 22. PMID 23176963
- [Background] Abensur Vuillaume L, Ferreira JP, Asseray N, Trombert-Paviot B, Montassier E, Legrand M, Girerd N, Boivin JM, Chouihed T, Rossignol P. Hypokalemia is frequent and has prognostic implications in stable patients attending the emergency department. PLoS One. 2020 Aug 4;15(8):e0236934. doi: 10.1371/journal.pone.0236934. eCollection 2020. PMID 32750075
- [Background] Ookuma T, Miyasho K, Kashitani N, Beika N, Ishibashi N, Yamashita T, Ujike Y. The clinical relevance of plasma potassium abnormalities on admission in trauma patients: a retrospective observational study. J Intensive Care. 2015 Aug 13;3(1):37. doi: 10.1186/s40560-015-0103-6. eCollection 2015. PMID 26269745
- [Background] Fleet JL, Shariff SZ, Gandhi S, Weir MA, Jain AK, Garg AX. Validity of the International Classification of Diseases 10th revision code for hyperkalaemia in elderly patients at presentation to an emergency department and at hospital admission. BMJ Open. 2012 Dec 28;2(6):e002011. doi: 10.1136/bmjopen-2012-002011. Print 2012. PMID 23274674
- [Background] Muschart X, Boulouffe C, Jamart J, Nougon G, Gerard V, de Canniere L, Vanpee D. A determination of the current causes of hyperkalaemia and whether they have changed over the past 25 years. Acta Clin Belg. 2014 Aug;69(4):280-4. doi: 10.1179/0001551214Z.00000000077. Epub 2014 Jun 18. PMID 24942977